CLINICAL TRIAL: NCT03748160
Title: Herd Immunity Communication and Influenza Vaccine Uptake
Brief Title: Herd Immunity and Influenza Vaccine Uptake
Acronym: HIIVU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: RWTH Aachen University (Other); University of Erfurt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 240317
Record Dates: First submitted 2018-11-01; First posted 2018-11-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — College Fraternities and Sororities

STUDY DESIGN:
Intervention Model Description: Cluster (household) RCT with three treatment arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): There is no intervention (letter) in the control arm. There is no control arm in the city of Espoo. 1/3 of subjects in all other municipalities are assigned to the control arm.
- Mailing (Active Comparator): This treatment arm consists of a standard letter reminding elderly citizens (65 years and above) about influenza vaccines that are available free of charge from the local health centers.
  Interventions: Other: Letter
- Herd (Active Comparator): This treatment arm consists of a letter that highlights the herd immunity effects of vaccination and reminds elderly citizens (65 years and above) about influenza vaccines that are available free of charge from the local health centers.
  Interventions: Other: Letter

INTERVENTIONS:
Other: Letter — Intervention consists of two different types of postal letters reminding elderly citizens (65 years and above) about influenza vaccines that are available free of charge from the local health centers
  Arms: Herd; Mailing

SUMMARY:
The aim of this study is to test the effectiveness of communicating the concept of herd immunity on actual influenza vaccine uptake using a randomized controlled trial.

DETAILED DESCRIPTION:
The investigators run a large-scale randomized controlled trial (RCT) to understand behavioural processes that guide decisions to vaccinate and test alternative strategies to communicate the concept of herd immunity. The experiment varies the text of postal letters send to individuals eligible for free influenza vaccines. The experiment is run in collaboration with the municipal health authorities.

The investigators identify from the Population Register all individuals who are born in year 1953 or before and resided in the participating municipality on October 01, 2018. The investigators will obtain the postal addresses of these individuals using the Population Register and randomly assign individuals to treatment conditions that differ in the wording of the information material and reception of a text message. Importantly, the extract from the Population Register will also include an individual identifier (social security number) that can be used to match the received type of letter (treatment) with the actual vaccination decision recorded in the Care Register for Health Care to objectively evaluate the impact of received information on vaccine uptake. The matching of postal addresses and vaccination data will be conducted using pseudonymized identifiers. The pseudonymization of individual identifiers will be performed separately for both datasets by professional data management and data security staff of the National Institute for Health and Welfare. The investigators conducting the data analysis will be able to access only pseudonymous data without a possibility to directly identify individuals from the data set. The data will be stored according to the data protection legislation and regulations of the National Institute for Health and Welfare during the research project.

The investigators randomly assign individuals to treatment conditions that differ in the wording of the letters. The authority's standard letter serves as the baseline condition (T1). This letter is extended by communicating the concept of herd immunity and appealing to pro-social preferences by highlighting the fact that vaccinations may effectively prevent infections among people who are not able to vaccinate themselves (especially babies) (T2). To summarize, this study includes a control treatment (T0, no letter) and two active treatment arms with the following contents:

T1 (Mailing) - Standard letter T2 (Herd) - Herd immunity letter

ELIGIBILITY:
Inclusion Criteria:

* At least 65 year old citizens in the municipalities of Espoo, Maalahti, Korsnäs, Kristiinankaupunki, Kaskinen and Närpiö

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48125 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Vaccine uptake | up to six months (beginning from November 1 / until April 30)
  Number of influenza vaccinations in study population

OTHER OUTCOMES:
Heterogeneity | up to six months (beginning from November 1 / until April 30)
  We run the statistical analysis by municipality to study ATE in areas with low/high historical vaccine uptake

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Betsch, PhD, Principal Investigator — University of Erfurt; Robert Böhm, PhD, Principal Investigator — RTWH Aachen University; Hanna Nohynek, PhD, Principal Investigator — Finnish Institute for Health and Welfare; Saila Pitkänen, MSc, Principal Investigator — Finnish Institute for Health and Welfare; Heini Salo, PhD, Principal Investigator — Finnish Institute for Health and Welfare; Lauri Sääksvuori, PhD, Study Director — Finnish Institute for Health and Welfare; Jonas Sivelä, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Health and Welfare, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided
This study is based in administrative register follow-up. We will share pseudonymized data according to current data availability regulations.

REFERENCES:
- [Derived] Saaksvuori L, Betsch C, Nohynek H, Salo H, Sivela J, Bohm R. Information nudges for influenza vaccination: Evidence from a large-scale cluster-randomized controlled trial in Finland. PLoS Med. 2022 Feb 9;19(2):e1003919. doi: 10.1371/journal.pmed.1003919. eCollection 2022 Feb. PMID 35139082